CLINICAL TRIAL: NCT00999817
Title: An Open Label Phase 1, Randomized Cross Over Trial To Estimate The Effect Of PF- 00299804 On The Pharmacokinetics Of Dextromethorphan In Healthy Volunteers
Brief Title: A Pharmacokinetic (PK) Study Of PF-00299804 And Dextromethorphan In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A7471039
Record Dates: First submitted 2009-10-08; First posted 2009-10-22 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Healthy Volunteers
Keywords: Drug-Drug interaction Study CYP2D6 inhibition Healthy Subjects
MeSH Terms: interventions — Dextromethorphan; dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Single 30 mg dose of dextromethorphan
  Interventions: Drug: reference [dextromethorphan]
- B (Experimental): Single 45 mg dose of PF-00299804 plus a single 30 mg oral dose of dextromethorphan
  Interventions: Drug: test [PF-00299804 + dextromethorphan]

INTERVENTIONS:
Drug: reference [dextromethorphan] — single 30 mg oral dose
  Arms: A
Drug: test [PF-00299804 + dextromethorphan] — single 45 mg oral dose of PF-00299804 and a single 30 mg oral dose of dextromethorphan
  Arms: B

SUMMARY:
A study to study the potential effect of PF-00299804 inhibition of CYP2D6 on dextromethorphan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non childbearing potential subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Subjects must be CYP2D6 extensive metabolizers, ultrarapid metabolizers or intermediate metabolizers, as predicted by CYP2D6 genotyping.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for men (1 drink =5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half lives preceding the first dose of study medication.
* 12 lead ECG demonstrating QTc >450 msec at Screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication. Depo Provera® must be discontinued at least 6 months prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of <1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results the study may be permitted on a case by case basis.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Plasma AUCinf, AUClast and Cmax of dextromethorphan and dextrorphan when given alone and when given in combination with PF- 00299804. | 7 weeks

SECONDARY OUTCOMES:
Plasma Tmax, t1/2, for dextromethorphan and dextrorphan and CL/F, and V/F for dextromethorphan (as data permit). | 7 weeks
Plasma AUCinf, AUClast, Cmax, Tmax, t1/2, CL/F, and V/F (as data permit) of PF 00299804 when given alone. | 7 weeks
Safety laboratory tests, physical examination, concomitant medication and adverse event monitoring. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471039&StudyName=A%20Pharmacokinetic%20%28PK%29%20Study%20Of%20PF-00299804%20And%20Dextromethorphan%20In%20Healthy%20Volunteers